CLINICAL TRIAL: NCT00840346
Title: A Phase I/II Multicenter, National, Open-Label Study of Panobinostat in Combination With Idarubicin and Cytarabine in Patients Aged 65 Years or Older With Newly Diagnosed Acute Myeloblastic Leukaemia (AML)
Brief Title: Panobinostat in Combination With Idarubicin and Cytarabine in Patients Aged 65 Years or Older With Newly Diagnosed Acute Myeloblastic Leukaemia (AML)
Acronym: PANOBIDARA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Josep Mª Ribera/Executive Secretary, PETHEMA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANOBIDARA
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Acute Myeloblastic Leukaemia
Keywords: Acute Myeloblastic Leukaemia (AML); Panobinostat
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The first patients enrolled in the trial will be successively distributed into three cohorts of patients for each dose level of panobinostat (20 mg, 30 mg, 40 mg) in combination with idarubicin and cytarabine, according to the classical 3+3 schedule
  Interventions: Drug: panobinostat

INTERVENTIONS:
Drug: panobinostat — 20 mg, 30 mg, 40 mg in combination with idarubicin and cytarabine, according to the classical 3+3 schedule.

SUMMARY:
This protocol is a multicenter, national, open-label, single-arm, non-controlled study designed to establish the efficacy (in terms of response and survival) and safety of panobinostat in combination with idarubicin and cytarabine and in monotherapy in patients with newly-diagnosed AML aged 65 years or older.

DETAILED DESCRIPTION:
A phase Ib will be initially performed to establish the MTD of panobinostat that can be administered in combination with the classic regimen of idarubicin and cytarabine in patients aged 65 years or older. This MTD will be established in the induction cycle. For this purpose, the first patients enrolled in the trial will be successively distributed into three cohorts of patients for each dose level of panobinostat (20 mg, 30 mg, 40 mg) in combination with idarubicin and cytarabine, according to the classical 3+3 schedule (vid section 5.2). In case of an unacceptable toxicity in the first dose step (20 mg), a dose reduction to a -1 step will be considered (10 mg). Patients included in the phase Ib part of the study will continue throughout the treatment with the starting dose of panobinostat corresponding to the step to which they were initially assigned (except for those patients receiving a dose higher than the MTD which will be deescalated to the MTD). 9 additional patients will be included at the MTD dose level to confirm the safety of this dose.

Once the MTD of panobinostat is determined, during the phase II of the study, up to a total of 46 patients will be recruited (40 of them at the MTD dose) and the scheduled assessments and visits will be carried out in three periods: Pre-treatment, Treatment, and Follow-up.

The pre-treatment period includes the screening visit where the written informed consent for participating in the study is obtained. Then, during the screening visit that is completed 14 days before the baseline visit (Days -14 to -1), patients are assessed for eligibility. The patients eligible for inclusion in the study will start the treatment period where they will receive two or three cycles of cytarabine and idarubicin in combination with panobinostat (induction and consolidation, or induction, re-induction and consolidation) followed by treatment with panobinostat as monotherapy (vid. schema in appendix 4). The induction cycle will comprise of cytarabine 100 mg/m2 (Day 1 to 7) and idarubicin 8 mg/m2 (Days 1 to 3) followed by panobinostat administered three times a week for three weeks (Days 8, 10, 12, 15, 17, 19, 22, 24, 26) (Table 4 ). The patients will be assessed by bone marrow aspiration on day +14 and at the moment of the recovery from aplasia.

If the patient experiences an unsatisfactory response, i.e. partial remission or resistant disease after the first cycle, a second induction cycle, identical to the first one (re-induction cycle), will be administered not sooner than seven days after receiving the last dose of panobinostat (in the induction cycle).

If the patient reaches a complete morphological remission (or CRi) after the induction or the re-induction cycles, then, in the absence of unacceptable toxicity, a consolidation cycle, identical to the induction cycle, will be administered once recovered from aplasia and always leaving the seven days of Panobinostat treatment free interval. If a patient does not reach a CR or CRi after the re-induction, she/he will be removed from the protocol.

Then, after the recovery from the aplasia caused by the last consolidation, all patients will be assessed for efficacy and safety, and, in the absence of relapse (i.e. patients in CR or CRi) or unacceptable toxicity will turn to the maintenance phase, during which they will receive single agent panobinostat at a dose of 40 mg with the following treatment regimen: three times a week for a total duration of three weeks (Days 1, 3, 5, 8, 10, 12, 15, 17 and 19), followed by a rest period of 9 days (Table 5). This cycle will be repeated every 28 days and a total of six cycles will be administered in the absence of relapse or unacceptable toxicity. During this period, patients will be assessed monthly for efficacy based on the hematimetric values (bone marrow aspirate will be performed every three months and when relapse is suspected) and toxicity/vital signs until the end of treatment.

Finally, during the follow-up period that starts once the patient completes the treatment, patients will be assessed for efficacy based on the hematimetric values (bone marrow aspirate will be performed every six months and when relapse is suspected) and toxicity every 3 months for one additional year.

Safety will be assessed by monitoring all adverse events, physical examination, vital signs, cardiological examinations, and blood and biochemical tests. The left ventricular ejection fraction (LVEF) will be assessed by echocardiography. The response to treatment will be assessed according to the standard Cheson response criteria. Furthermore, the impact of MRD in the prognosis of these patients will be assessed. For this purpose, MRD changes at different treatment time points will be tested by multiparametric flow cytometry: at Day +14 post-induction, before starting the first consolidation cycle (this is to say at the moment of achieving CR), at the start of maintenance therapy, every three months during this phase and every six months during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The patient should, in the investigator's opinion, be able to meet all clinical trial requirements.
* The patient should have voluntarily give the informed consent before performing any study test that is not part of the regular care of the patients.
* Age > 65 years.
* The patient should be diagnosed with AML according to the standard criteria of the World Health Organisation (WHO) (see Appendix 8).
* The patient should not have received any prior treatment for AML.
* The patient should have a performance status measured by the ECOG scale <= 2 .
* The patient should have the following laboratory values prior to the start of the treatment:

  * Aspartate transaminase (AST): ≤ 2.5 x the upper normal ranges.
  * Alanine transaminase (ALT): ≤ 2.5 x the upper normal ranges.
  * Total bilirubin: ≤ 1.5 x the upper normal ranges.
  * Alkaline phosphatase: ≤ 2.5 x the upper normal ranges.
  * Serum creatinine ≤ 2 mg/dl.
  * Serum potassium, magnesium, phosphorus, sodium, total calcium (corrected for serum albumin) or ionized calcium within normal limits (WNL) for the institution. Note: Electrolytes (supplemental therapy) should be given to correct values that are <LLN. Post-correction values must not be deemed to be a clinically significant abnormality prior to patients being dosed.
* Left ventricular ejection fraction measured by echocardiography ≥ 50%

Exclusion Criteria:

* Patients previously receiving treatment with histone deacetylase inhibitors (HDACi).
* Patient will need valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat dose.
* Promyelocytic AML (M3).
* Secondary AML or previous history of MDS.
* Male patients whose sexual partners are women of a fertile age and do not use contraceptive.
* Known brain or leptomeningeal involvement.
* Presence of any limitation affecting the ability of the patient to comply with the treatment.
* Patients receiving any investigational agent in the 30 days prior to inclusion.
* Patient carrier of human immunodeficiency virus (HIV), hepatitis B virus surface antigen or active infection by hepatitis C virus.
* Presence of heart disorders or clinically significant heart diseases, including any of the following:

  * Congenital QT prolongation "long QT syndrome").
  * History or presence of sustained ventricular tachyarrhythmia (patients with a history of atrial arrhythmia are acceptable, but this must be discussed with the sponsor prior to inclusion).
  * Any history of ventricular fibrillation or "torsade de pointes".
  * Bradycardia defined as HR < 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
  * Screening ECG with QTc > 450 msec.
  * Right bundle branch block + left anterior hemiblock (bifascicular block).
  * Patients with acute myocardial infarction or unstable angina ≤ 6 months before the start of the investigational drug.
  * Any clinically significant heart disease (e.g., NYHA grades III or IV, or baseline LVEF <45%, uncontrolled hypertension, or history of poor compliance of antihypertensive treatment).
* Gastrointestinal disease making panobinostat absorption significantly difficult.
* Diarrhea > grade 1 according to CTCAE criteria, version 3.0.
* Any serious or uncontrolled medical condition (e.g., uncontrolled diabetes, or active or uncontrolled infection), including laboratory disorders that could involve unacceptable risks or affect protocol compliance.
* Concomitant administration of drugs with a relative risk of increasing the QT interval or inducing "torsade de pointes" if this treatment cannot be discontinued or replaced by another prior to the start of the test drug.
* Patient has active bleeding diathesis or is currently being treated with therapeutic doses of sodium warfarin (Coumadin®) or other vitamin K active agents Note: mini-dose of Coumadin® (e.g., 1 mg/day) or anti-coagulants given to maintain intravenous line patency, as well as unfractionated or low molecular weight heparin therapy is permitted
* Patients undergoing major surgery in the four weeks prior to the start of the study treatment or not recovering from the treatment adverse events.
* Patients with a history of malignancies in the past five years. Basal cell carcinoma, skin epithelioma and carcinoma of the cervix in situ are excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of panobinostat in combination with idarubicin and cytarabine after an induction cycle in patients aged 65 years or older with newly diagnosed AML | 1 year
To analyse efficacy in terms of response to an induction (+/- reinduction) and consolidation regimens with idarubicin and cytarabine in combination with panobinostat | 2 years
To explore efficacy in terms of TTR during a maintenance period with panobinostat as monotherapy in patients aged 65 years or older with newly diagnosed AML | 2 years

SECONDARY OUTCOMES:
Investigation of the overall safety and tolerability of panobinostat when given in combination with idarubicin and cytarabine, with special focus on cardiac safety determined by echocardiography and ECG monitoring | 1 year
Survival: Overall survival, disease-free survival, and duration of response | 4 years
Impact of Panobinostat in the reduction of the minimum residual disease (MRD) monitored by multiparametric flow cytometry at different time points of the study: During the induction and consolidation treatments and during the maintenance treatment | 4 years
To investigate the safety and tolerability of panobinostat in combination with idarubicin and cytarabine and of panobinostat as monotherapy measured in terms of incidence of clinical and biological toxicity | 2 years

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital Germans Trías i Pujol, Barcelona
  - Hospital Santa Creu y Sant Pau. Barcelona, Barcelona
  - Hospital 12 de Octubre. Madrid, Madrid
  - Hospital Clínico San Carlos. Madrid, Madrid
  - Hospital Ramón y Cajal. Madrid, Madrid
  - Hospital Morales Messeguer. Murcia, Murcia
  - Hospital Univ. La Fe de Valencia, Valencia
  - Hospital Lozano Blesa. Zaragoza, Zaragoza

REFERENCES:
- [Derived] Ocio EM, Herrera P, Olave MT, Castro N, Perez-Simon JA, Brunet S, Oriol A, Mateo M, Sanz MA, Lopez J, Montesinos P, Chillon MC, Prieto-Conde MI, Diez-Campelo M, Gonzalez M, Vidriales MB, Mateos MV, San Miguel JF; PETHEMA Group. Panobinostat as part of induction and maintenance for elderly patients with newly diagnosed acute myeloid leukemia: phase Ib/II panobidara study. Haematologica. 2015 Oct;100(10):1294-300. doi: 10.3324/haematol.2015.129577. Epub 2015 Jul 9. PMID 26160880
- See also: Spanish Association of Hematology — http://aehh.org
- See also: CRO — http://dynasolutions.com